CLINICAL TRIAL: NCT00950469
Title: Comparison of the New High Sensitive Cardiac Troponin T With the 4th Generation Troponin-T, Myoglobin, Heart-type Fatty Acid Binding Protein for Early Identification of Myocardial Necrosis in Patients With Suspected Acute Coronary Syndrome
Brief Title: TnThs for Identification Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: Prof. Dr. Evangelos Giannitsis (Unknown)
Responsible Party: Prof. Dr. Evangelos Giannitsis, University of Heidelberg
Other Study IDs: TnThs 1
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Acute Coronary Syndrome
Keywords: high sensitive troponin T; cardiac necrosis; early detection; myoglobin; h-FABP; early identification and risk stratification of patients with suspicious acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum) were collected at presentation and after 6 hours. After collection, serum was centrifuged immediately and stored at -80°C until analysis.
  The laboratory staff responsible for measurements was blinded to patient data.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with acute coronary syndrome: 94 consecutive patients without ST-segment elevation admitted to the Chest Pain Unit of the University of Heidelberg were enrolled with symptoms suggestive of ACS.
  Unstable angina and non-ST-segment elevation myocardial infarction were diagnosed using the joint European Society of Cardiology/American College of Cardiology/American Heart Association/World Heart Federation Task Force redefinition of myocardial infarction guidelines. Patients with ST-segment elevation were excluded.

SUMMARY:
OBJECTIVES/BACKGROUND: We sought to determine the early diagnostic value of the new high sensitive cardiac troponin T assay (TnThs) in suspected acute coronary syndrome (ACS) and to compare it with the 4th generation cTnT assay from the same manufacturer, myoglobin and heart-type fatty acid binding protein (h-FABP).

METHODS: The study consisted of 94 patients with chest pain admitted to the chest pain unit with the diagnosis of suspected ACS without ST-Elevation. Patients were divided according to time from onset of symptoms to presentation into an early presenter group (<4 hours) and a late presenter group (≥4 hours).

A median of 6 samples (range 2-8) were available per patient. The diagnostic performance of TnThs was assessed using ROC analysis and areas under the curve (AUC) of baseline and follow-up results of TnThs, cTnT, myoglobin, and h-FABP were compared using c-statistics.

RESULTS: The TnThs assay allows an excellent prediction of non-ST-segment-elevation myocardial infarction (non-STEMI) at presentation.A follow-up sample improves diagnostic performance in a time dependent manner. The AUC of the TnThs was superior to cTnT at all time points.

CONCLUSIONS: A baseline sample of TnThs allows an earlier prediction of non-STEMI than the less sensitive and precise 4th generation cTnT assay. The excellent performance of TnThs at baseline and follow-up might obviate the need for other early necrosis markers.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with ACS

Exclusion Criteria:

* Patients with ST-segment elevation at presentation were excluded as were patients with muscular trauma, or severe kidney dysfunction defined as an estimated glomerular filtration rate below 60 ml/min/1.73m2.
* In addition patients who underwent percutaneous coronary intervention during follow-up sampling were also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 94 consecutive patients without ST-segment elevation admitted to the Chest Pain Unit of the University of Heidelberg were enrolled with symptoms suggestive of ACS.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the early diagnostic value of the new high sensitive cardiac troponin T assay (TnThs) for earlier detection of myocardial necrosis in suspected acute coronary syndrome. | 6 to 24 hours after admission

SECONDARY OUTCOMES:
Comparison of TnThs with cTnT, myoglobin and h-FABP. | 6 to 24 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, MD, FACC, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany